CLINICAL TRIAL: NCT03802747
Title: Phase I Study of Dual Immune Checkpoint Blockade (Anti-PD-L1 (Durvalumab) (MEDI4736) and Anti-CTLA4 (Tremelimumab) Plus Yttrium-90 (Y-90) Radioembolization & Stereotactic Body Radiation Therapy (SBRT) in Refractory Metastatic MSS (Microsatellite Stable) Colorectal Cancer With Liver Metastases
Brief Title: Immunotherapy Combined With Y-90 and SBRT for Colorectal Liver Metastases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Colorado, Denver (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0710.cc; ESR-17-13132 (Other: Astra Zeneca)
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: Liver Metastases; Phase 1; Durvalumab; Tremelimumab; Yttrium-90; Radioembolization; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; tremelimumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: The first 6 patients will receive durvalumab alone with Y-90 and SBRT followed by 4 months of durvalumab. The next 6 patients will received durvalumab with Y-90 and SBRT followed by 4 months of durvalumab + tremelimumab.Durvalumab will be dosed at 1500 mg fixed dosing every 4 weeks and continued at this interval until progression or dose-limiting toxicity. There will be no dose escalation. For patients who will receive both Durvalumab and Tremelimumab, the Tremelimumab will be dosed at 75 mg every 4 weeks (same day as durvalumab infusion) for a maximum of 4 doses. There will be no dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Y-90, SBRT, and Durvalumab Alone (Experimental): Six patients will be enrolled in cohorts of three to be administered Y-90, SBRT, and Druvalumab.
  Interventions: Drug: Durvalumab; Drug: Y-90 Selective Internal Radiation Therapy (SIRT); Drug: Stereotactic Body Radiation Therapy (SBRT)
- Y-90, SBRT, and Durvalumab + Tremelimumab (Experimental): Six patients will be enrolled in cohorts of three to be administered Y-90, SBRT, and Druvalumab + Tremelimumab.
  Interventions: Drug: Durvalumab and Tremelimumab; Drug: Y-90 Selective Internal Radiation Therapy (SIRT); Drug: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be dosed at 1500 mg fixed dosing every 4 weeks and continued at this interval until progression or dose-limiting toxicity.
  Arms: Y-90, SBRT, and Durvalumab Alone
Drug: Durvalumab and Tremelimumab — Durvalumab will be dosed at 1500 mg fixed dosing every 4 weeks and continued at this interval until progression or dose-limiting toxicity. Tremelimumab will be dosed at 75 mg every 4 weeks (same day as durvalumab infusion) for a maximum of 4 doses.
  Arms: Y-90, SBRT, and Durvalumab + Tremelimumab
Drug: Y-90 Selective Internal Radiation Therapy (SIRT) — Yttrium-90 microsphere therapy consists of resin beads loaded with Yttrium, a pure beta emitter with a 64.2 hour half-life. Radioembolization will be performed as standard of care therapy per current NCCN guidelines.
Drug: Stereotactic Body Radiation Therapy (SBRT) — High-dose hypofractionated conformal external beam radiation therapy that is considered a standard of care. SBRT will also be considered for metastases that are persistent and/or progressive after Y-90 based on MR imaging and pathology from tissue biopsies.

SUMMARY:
This study is evaluating the combination of Y-90 radioembolization followed by SBRT with the immunotherapy drugs, durvalumab and tremelimumab, to improve disease control of liver metastases for patients with microsatellite stable colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic confirmation of metastatic microsatellite stable colorectal cancer
2. Liver metastases not amenable to resection for which palliative Y-90 and SBRT is considered appropriate standard therapy
3. Patients should have received at least one prior standard therapy for metastatic disease. Prior therapies should include regimens containing oxaliplatin and irinotecan in combination with a fluoropyrimidine if appropriate (e.g., FOLFOX and FOLFIRI or their variants) unless contraindicated, not tolerated, or declined.
4. Male or female, age 18 or older
5. ECOG performance status of 0 or 1
6. Body weight >30 kg
7. Life expectancy of greater than 6 months
8. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Patients must have acceptable organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC ≥1.0 x (> 1000 per mm3))
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
   * Total bilirubin : < 2x upper limit of normal
   * AST (SGOT)/ALT (SGPT): <2.5x institutional upper limit of normal
   * Creatinine: <1.5x upper limit of normal OR Creatinine clearance >40mL/min for patients with creatinine levels above institutional normal
10. Ability to understand and willingness to sign a written informed consent document
11. Residual or on-going ≥ Grade 3 treatment-related toxicity from previous chemotherapy should be resolved.

Exclusion Criteria:

1. Participation in another clinical study with an investigational drug during the last 4 weeks.
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade >2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
6. History of allogenic organ transplantation.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
8. Prior therapy with an anti-PD-1 or anti-PD-L1, including durvalumab antibody within 6 months prior to enrollment and anti-CTLA4 (including tremelimumab)
9. Prior abdominal radiotherapy
10. Child-Pugh class B or higher
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, insterstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis
14. History of active primary immunodeficiency
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Contraindication to IV contrast
19. Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy are excluded. This applies to any woman who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH levels greater than 35 mIU/mL). A negative urine or serum pregnancy test must be obtained within 14 days prior to the start of study therapy in all women of child-bearing potential. Male subjects must also agree to use effective contraception for the same time period as above.
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
21. Use of any prohibited concomitant medications, including:

    * Traditional herbal medicines, as their use may result in unanticipated drug-drug interactions that may cause or confound assessment of toxicity.
    * Any live, attenuated vaccine (e.g., FluMist) within 4 weeks prior to Cycle 1 Day 1 or at any time during the study and for at least 5 months after the last dose of durvalumab.
    * Use of steroids to premedicate patients for whom MRI scans with contrast are contraindicated (i.e., patients with contrast allergy or impaired renal clearance)
    * Immunomodulatory agents, including but not limited to interferons or interleukin-2, during the entire study; these agents could potentially increase the risk for autoimmune conditions when administered with durvalumab.
    * Immunosuppressive medications, including but not limited to cyclophosphamide, azathioprine, methotrexate, and thalidomide; these agents could potentially alter the activity and the safety of durvalumab
    * Systemic corticosteroids and tumor necrosis factor-α (TNF-α) inhibitors may attenuate potential beneficial immunologic effects of treatment with durvalumab. Therefore, in situations where systemic corticosteroids or TNF-α inhibitors would be routinely administered, alternatives, including antihistamines, should be considered first by the treating physician. If the alternatives are not feasible, systemic corticosteroids and TNF-α inhibitors may be administered at the discretion of the treating physician (see Section 4.4.2)
    * Initiation or increased dose of granulocyte colony-stimulating factors (e.g., granulocyte colony stimulating factor, granulocyte/macrophage colony-stimulating factor, and/or pegfilgrastim) is prohibited.
22. Shunt Fraction greater than 20% (Requires more than 30gy dose to the lungs in order receive therapeutic dose of Y-90).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related Adverse Events | Start of study to 3 months post treatment completion, up to 5 years
  Adverse events related to Y-90, SBRT, and durvalumab plus tremelimumab will be summarized by dose and severity as assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Dose-Limiting Toxicity of Y-90+SBRT in Combination with Dual Immune Checkpoint Blockade | Start of study to 3 months post treatment completion, up to 5 years
  Defined as the rate of >Grade 3 treatment-related adverse events during treatment or within 3 months of treatment completion.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  The determination of antitumor activity will be based on objective response assessments as defined by RECIST version 1.1 and immune RECIST.
Progression Free Survival for Three Months (PFS) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  The determination of antitumor activity will be based on objective response assessments as defined by RECIST version 1.1 and immune RECIST.
Overall Response Rate (ORR) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  The determination of antitumor activity will be based on objective response assessments as defined by RECIST version 1.1 and immune RECIST.
Overall Survival for Two Years (OS) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  Measure of overall survival rate by examining the incidence of death over a two year period.
Liver Progression Free Survival for One Year (L-PFS) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  The determination of antitumor activity will be based on objective response assessments as defined by RECIST version 1.1 and immune RECIST.
Pathological Response Rates (PRR) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  Measured by the percentage of viable tumor throughout and post treatment
Time to Tumor Progression (TTP) | Landmark time of initiation of tremelimumab, about 18 weeks after the start of treatment, to end of follow up, up to 2 years
  The determination of antitumor activity will be based on objective response assessments as defined by RECIST version 1.1 and immune RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Karyn Goodman, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No